CLINICAL TRIAL: NCT02008994
Title: A Phase II Pilot Study Utilizing Genomic and Proteomic Profiling to Find Potential Targets and Influence Treatments for Patients With Metastatic Breast Cancer
Brief Title: Phase II Study Using Genomic & Proteomic Profiling to Influence Treatments for Patients With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Resignation of Principal Investigator
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SH SSKT001
Record Dates: First submitted 2013-10-30; First posted 2013-12-11 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer; breast cancer; genomics; personalized medicine; precision oncology; breast cancer treatment; metastatic breast cancer treatment; genetic testing and breast cancer treatment; breast cancer trial; metastatic breast cancer trial
MeSH Terms: conditions — Breast Neoplasms | interventions — Genome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Genomic and Proteomic Profiling (Experimental): * Reverse Phase Protein Microarray will be used to determine how often there are specific proteins that could make your tumor susceptible or resistant to treatment.
  * Immunohistochemistry will look for specific markers of disease in your DNA.
  * RNA sequencing will be used to help doctors and scientists understand how your genes are working.
  * Low pass whole genome and exome sequencing will be used to help identify variants in your DNA.
  Interventions: Other: Genomic and Proteomic Profiling

INTERVENTIONS:
Other: Genomic and Proteomic Profiling — Following review of targets by the Treatment Selection Committee, the treating physician will decide whether to continue with planned therapy or alter the course of treatment based on the genomic results.

SUMMARY:
Genes are the basic "instruction book" for the cells that make up our bodies and are made out of DNA. Many research studies are done to find the best possible way to treat patients with cancer. Recently there has been a great deal of interest in developing new anticancer agents that are more targeted to a patient's individual genetic information, as well as diseases caused by defects in a person's genes.

Identification of precisely which treatments to use against a specific patient's tumor is challenging. In this study, four cutting-edge technologies will be used to identify genomic (information we get from DNA and RNA) and proteomic (information we get from proteins) targets for the treatment of your tumor. These four tests will be used together to gather information about your tumor giving doctors and scientists a better understanding of the structure of your tumor and what the best treatment or combination of treatments may be for you. The therapy you receive to treat your tumor will be based on your medical history, previous treatments for your disease if applicable, current state of health, and the findings from these four tests. The therapy you ultimately receive will be selected by your doctor in consultation with a panel of experts in cancer and cancer genomics (the Treatment Selection Committee).

DETAILED DESCRIPTION:
DNA contains genetic information that acts as a blueprint for how parts of your body are made and work, determining such things as eye and hair color. DNA is made up of long strands of repeating letters that form a code. The order in which these letters are written is very precise. In the same way that a spelling mistake in a word could change its meaning entirely (for example, mean and meat), a single change in the sequence of DNA can lead to a change in how the body works, which may lead to disease. Currently, researchers and doctors know some of the genetic changes that may result in disease, but they do not know all of the genetic changes that can cause disease.

Proteins are the basic building blocks of your body. The parts of your body such as your muscles, your skin, and your organs are made up mostly of proteins. DNA provides the plans, or instructions, for how each protein should be made. If there is a change in your DNA, there may be a change in how a protein is made. Sometimes these changes can lead to disease. To make a protein, the cells in your body take the DNA and make a copy called RNA. The cells read the RNA to make the protein. DNA can be thought of as the original master plan with RNA being photocopies of this plan. The number of copies of RNA can determine the amount of protein that can be made. If the body needs more protein, it can make more RNA but if it needs less protein, it can also shred the RNA so that it cannot be read. The amount of a particular RNA or protein can also be important in how the body works. Too much or too little of a particular protein can also lead to disease. Understanding the relationship between DNA, RNA and proteins can be important in knowing what causes disease and how to treat it.

Identification of precisely which treatments to use against a specific patient's tumor is challenging. In this study, four cutting-edge technologies will be used to identify genomic (information we get from DNA and RNA) and proteomic (information we get from proteins) targets for the treatment of your tumor. These four tests will be used together to gather information about your tumor giving doctors and scientists a better understanding of the structure of your tumor and what the best treatment or combination of treatments may be for you. The therapy you receive to treat your tumor will be based on your medical history, previous treatments for your disease if applicable, current state of health, and the findings from these four tests. The therapy you ultimately receive will be selected by your doctor in consultation with a panel of experts in cancer and cancer genomics (the Treatment Selection Committee).

The purpose of this study is to examine the impact of targeted therapy for breast cancer based upon proteomic and genomic profiling using four different methods of analysis.

* Reverse Phase Protein Microarray will be used to determine how often there are specific proteins that could make the tumor susceptible or resistant to treatment.
* Immunohistochemistry will look for specific markers of disease in DNA.
* RNA sequencing will be used to help doctors and scientists understand how genes are working.
* Low pass whole genome and exome sequencing will be used to help identify variants in DNA.

The goal of this study will be to enroll at least 25 women who will receive therapy influenced by the results derived from genomic and proteomic profiling. Up to 30 women will receive treatment suggested by an identified target and up to 10 women will receive treatment that the subject and her doctor choose. The actual treatment of disease will be based upon multiple factors, including current physical condition, prior therapies if applicable, standard labs and tests, and physician's preference. The results from the genomic and proteomic profiling will add to the available information that will be used to aid us in deciding upon the course of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Understand and provide written informed consent and HIPAA Authorization prior to initiation of any study-specific procedures
* Have a life expectancy of >3 months
* Have a diagnosis of metastatic breast cancer with measurable disease (RECIST 1.1)
* Have documentation of progression if applicable (by RECIST 1.1) on the treatment regimen immediately prior to entering this study.
* Be ≥ 18 years of age
* Have an ECOG score of 0-1
* Be a good medical candidate for and willing to undergo two biopsies or surgical procedures to obtain tissue, which may or may not be part of the patient's routine care for their malignancy. The 1st biopsy is required and the 2nd biopsy is optional.
* Have documented lack of response or documented progression form last therapy.
* Have adequate organ and bone marrow function as defined below:
* Bone marrow: absolute neutrophil count (ANC) ≥ 1.5 x 109/L; hemoglobin 9 g/dL; platelets > 100 x 109/L
* Renal: creatinine clearance ≥ 60 mL/min (calculated according to Cockcroft and Gault) or creatinine ≤ 1.5 mg/dL
* Hepatic: bilirubin ≤ 2.5 x the upper limit of normal (ULN); aspartate transaminases (AST/SGOT); alanine transaminases (ALT/SGPT) ≤ 2.5 x ULN (or ≤ 5 x ULN if due to underlying liver metastases); INR ≤ 1.5 x ULN (except in the case of anti-coagulation therapy)
* Female patients of childbearing potential must have a negative pregnancy test and agree to use at least one form of contraception during the study and for at least one month after treatment discontinuation. For the purposes of this study, child- bearing potential is defined as: all female patients that were not in post- menopause for at least one year or are surgically sterile
* Male patients must use a form of barrier contraception approved by the investigator / treating physician during the study and for at least one month after treatment discontinuation

Exclusion Criteria:

* Have a tumor biopsy intended for use in the current study that was performed more than 2 months prior to analysis
* Have metastatic lesions that are not accessible to biopsy
* Have had interventional cancer therapy conducted after the biopsy was collected prior to analysis
* Have symptomatic CNS metastasis. Patients with a history of CNS metastases who have been treated with whole brain irradiation must be stable without symptoms for 4 weeks after completion of treatment, with image documentation required, and must be either off steroids or on a stable dose of steroids for ≥ 2 weeks prior to enrollment
* Have any previous history of another malignancy (other than cured basal cell carcinoma of the skin or cured in-situ carcinoma of the cervix) within 5 years of study entry
* Have uncontrolled concurrent illness including, but not limited to, ongoing or active serious infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmias, psychiatric illness, or situations that would limit compliance with the study requirements or the ability to willingly give written informed consent
* Have known HIV, HBV, HCV infection
* Are pregnant or breast-feeding patients or any patient with childbearing potential not using adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival as a result of targeted therapy for breast cancer suggested by proteomic and genomic profiling using RPMA, targeted resequencing, IHC analysis, WGS, RNA-Seq, and Exome sequencing. | Disease status will be assessed every 7 ± 1 weeks until progression or time of treatment discontinuation, whichever is later.

SECONDARY OUTCOMES:
The frequency in which proteomic, IHC, and genomic profiling analysis of a tumor by RPMA, targeted resequencing, IHC analysis, WGS, RNA-Seq, and Exome sequencing yields a target. | Results of profiling will be made available to investigators within 10 working days of receipt of tissue specimens.
The frequency of changes to initial treatment recommendations after re-biopsy and analysis after 7 ± 2 days of treatment. | After 7 ± 2 days of treatment.
Results of LCM vs non-LCM samples on determination of driving mutations, transcripts, and alternative pathway activation. | Within one year after enrollment.
The percent of time in which RPMA, targeted resequencing, IHC analysis, RNA-Seq, and Exome sequencing based treatment is different than that which would have been selected by the patient's physician. | Within one year of study closing to enrollment.
Structural changes and copy number variants meaning after identification using low pass whole genome sequencing (WGS). | At initial biopsy and day 7 biopsy (if performed).
Response rate (according to RECIST 1.1 response criteria) - the percent of patients with non-progression at 4 months, and - overall survival, in patients whose therapy is selected by proteomic and genomic analysis and IHC analysis. | At 4 months.
Number of patients, as a whole, where the optimal tissue biomarker subset is most predictive of a given therapy leading to an improved outcome. | Within one year of closing to enrollment.
Physician and patient expectations, attitudes, experiences, and psychological responses to the use of proteomic and genomic profiling in breast cancer. | Within one year of closing to enrollment.
  A questionnaire will be provided to physicians and patients to measure their knowledge regarding genomics and the interaction with cancer care.
Patient symptoms identified by the Therapy-Related Symptom Checklist (TRSC) correlate with any associated SNPs identified through genomic analysis | Within one year of closing to enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: David Pearce, PhD, Study Director — Sanford Research
Locations (1):
- Sanford Health, Sioux Falls, South Dakota, United States